CLINICAL TRIAL: NCT00483665
Title: Detection of Endoleak by Vasovist-Enhanced Magnetic Resonance Imaging
Brief Title: Vasovist Endoleak Study
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: M. Prokop, UMC Utrecht
Other Study IDs: UMC_06_112
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: endoleak
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Computed tomography angiography — Computed tomography angiography
Procedure: Magnetic resonance imaging — Magnetic resonance imaging after injection of Vasovist

SUMMARY:
After endovascular treatment of an abdominal aortic aneurysm, lifelong imaging follow-up is needed to monitor the effectiveness of the treatment. One parameter in this follow-up is endoleak, which is leakage of blood into the aneurysm sac. The aim of this study is to investigate the value of magnetic resonance imaging using Vasovist as a contrast agent for the detection of endoleaks.

DETAILED DESCRIPTION:
After endovascular abdominal aortic aneurysm repair, life-long follow-up is needed to monitor the effectiveness of exclusion of the aneurysm sac from blood flow. For this reason, aneurysm diameter and the presence of endoleaks is evaluated with computed tomographic (CT) angiography yearly after Endovascular Aneurysm Repair (EVAR).

The aim of this study is to investigate the value of magnetic resonance imaging using Vasovist as a contrast agent for the detection of endoleaks.

The advantages of magnetic resonance imaging with respect to CTA are no use of ionizing radiation, use of less nephrotoxic contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* Patient is more than one year after endovascular abdominal aortic aneurysm repair
* Patient has a stable or growing aneurysm according to diameters measured on CT angiography images
* No evidence of endoleak on recent CT angiography

Exclusion Criteria:

* contraindication for MRI examination

  * claustrophobia
  * pacemaker
  * other non-MRI compatible implants
* contraindication for use of contrast agent

  * known allergy to drugs or contrast media
  * MRI examination with the use of gadolinium within 24 hours of the blood-pool agent injection
  * severe renal impairment = creatine > 2 mg/dl (=176 mmol/l)
  * patient clinically instable
  * Participation in drug research within 30 days before and 1 day after MRI-examination with use of Vasovist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients after more than 1 year who have a stable or growing aneurysm according to diameters measured on CT angiography images and no evidence of endoleak on recent CT angiography
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Prokop, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands